CLINICAL TRIAL: NCT07353281
Title: Carbetocin Versus Misoprostol for the Prevention of Postpartum Hemorrhage After Vaginal Delivery in Women With Risk Factors: A Prospective Randomized Study
Brief Title: Carbetocin vs Misoprostol for Postpartum Hemorrhage Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr Raneen Abu Shqara, Dr., Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0206-25-NHR
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Complication; Postpartum Hemorrhage
Keywords: Postpartum hemorrhage, Carbetocin, Misoprostol, Vaginal delivery, Uterotonic agents, High-risk pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Injections; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin arm (Experimental): Participants in this arm will receive intravenous carbetocin (100 micrograms) immediately after placental delivery for the prevention of postpartum hemorrhage following vaginal delivery. Carbetocin will be administered as part of active management of the third stage of labor in women at increased risk for postpartum hemorrhage.
  Interventions: Drug: Carbetocin 100 Microgram/mL Solution for Injection
- Misoprostol arm (Active Comparator): Participants in this arm will receive rectal misoprostol (1000 micrograms) immediately after placental delivery, in addition to intravenous oxytocin, for the prevention of postpartum hemorrhage following vaginal delivery. This regimen represents an accepted uterotonic prophylaxis strategy for women at increased risk for postpartum hemorrhage.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Carbetocin 100 Microgram/mL Solution for Injection — Participants randomized to this intervention will receive intravenous carbetocin 100 micrograms administered immediately after placental delivery as prophylaxis for postpartum hemorrhage following vaginal delivery. Carbetocin is a long-acting synthetic analogue of oxytocin and is used as part of active management of the third stage of labor in women at increased risk for postpartum hemorrhage.
  Arms: Carbetocin arm
Drug: Misoprostol — Participants randomized to this intervention will receive rectal misoprostol 1000 micrograms immediately after placental delivery for the prevention of postpartum hemorrhage following vaginal delivery. In accordance with standard practice, intravenous oxytocin 10 units will also be administered as part of active management of the third stage of labor in women at increased risk for postpartum hemorrhage.
  Arms: Misoprostol arm

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal morbidity and mortality worldwide, particularly among women with known risk factors. Uterotonic agents are routinely administered after vaginal delivery to prevent excessive bleeding. Carbetocin, a long-acting oxytocin analogue, and misoprostol are both used for this purpose, but comparative data in high-risk vaginal deliveries remain limited.

This prospective randomized study aims to compare the effectiveness and safety of intravenous carbetocin versus rectal misoprostol for the prevention of postpartum hemorrhage in women with risk factors undergoing vaginal delivery at Galilee Medical Center. The primary outcome is the incidence of postpartum hemorrhage. Secondary outcomes include the need for additional uterotonic agents or surgical interventions, changes in hemoglobin levels, blood transfusion requirements, and maternal adverse effects.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH), most commonly caused by uterine atony, remains a major contributor to maternal morbidity and mortality. Women with established risk factors-such as grand multiparity, prior PPH, prolonged labor, fetal macrosomia, polyhydramnios, chorioamnionitis, or prolonged oxytocin exposure-are at particularly increased risk following vaginal delivery.

Active management of the third stage of labor using uterotonic medications is the cornerstone of PPH prevention. Oxytocin is widely used but has a short half-life, often requiring repeated dosing or continuous infusion. Carbetocin is a synthetic oxytocin analogue with a longer half-life and sustained uterotonic effect, which may offer improved prophylaxis against PPH. Misoprostol, a prostaglandin E1 analogue, is also commonly used due to its low cost, ease of administration, and stability, although it is associated with gastrointestinal and thermoregulatory side effects.

While carbetocin has demonstrated superiority over oxytocin in cesarean deliveries, evidence comparing carbetocin with misoprostol in high-risk vaginal deliveries is limited. This prospective, randomized, single-center study will enroll women at term with singleton pregnancies and predefined risk factors for postpartum hemorrhage. Participants will be randomized in a 1:1 ratio to receive either intravenous carbetocin (100 µg) or rectal misoprostol (1000 µg) with standard oxytocin after placental delivery.

The primary outcome is the occurrence of postpartum hemorrhage. Secondary outcomes include the need for additional uterotonic agents, blood transfusion, uterine revision or manual placental removal, changes in hemoglobin levels before and after delivery, duration of maternal hospitalization, and maternal adverse effects such as diarrhea, shivering, headache, and facial flushing.

This study aims to provide high-quality prospective data to guide the optimal prophylactic uterotonic strategy for women at increased risk of postpartum hemorrhage following vaginal delivery.

ELIGIBILITY:
Inclusion Criteria

* Women aged 18 years or older
* Singleton pregnancy
* Gestational age 37-42 weeks
* Cephalic presentation
* Vaginal delivery
* Presence of one or more risk factors for postpartum hemorrhage, including:
* Grand multiparity (≥5 previous deliveries)
* History of postpartum hemorrhage
* History of manual removal of placenta
* Estimated fetal weight ≥4,000 grams
* Polyhydramnios
* Chorioamnionitis
* Prolonged oxytocin use during labor (third augmentation cycle or more)
* Eligible for prophylactic uterotonic therapy after delivery
* Provided written informed consent

Exclusion Criteria

* Multiple gestation
* Known major fetal anomalies
* Intrauterine fetal demise (IUFD)
* Contraindication to vaginal delivery
* Known hypersensitivity to carbetocin, misoprostol, or oxytocin
* Known coagulation disorders requiring alternative management
* Planned cesarean delivery
* Participation in another interventional study that may affect postpartum bleeding outcomes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is limited to pregnant women.
Enrollment: 146 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum hemorrhage (PPH) | Within 24 hours after delivery
  Postpartum hemorrhage defined as estimated blood loss ≥1,000 mL within 24 hours after vaginal delivery, or any bleeding associated with hemodynamic instability requiring medical or surgical intervention, according to institutional protocol.
Need for additional uterotonic treatment or surgical intervention | Within 24 hours of delivery
  Requirement for additional uterotonic agents (including oxytocin infusion, methylergonovine, carboprost, or misoprostol), uterine massage, uterine revision, or surgical intervention for management of postpartum bleeding.

SECONDARY OUTCOMES:
Change in hemoglobin level | From admission to 24-48 hours postpartum
  Difference between pre-delivery and post-delivery hemoglobin concentration, measured in g/dL.
Blood transfusion requirement | Up to 24-48 hours postpartum
  Administration of packed red blood cells or other blood products during or after delivery.
Maternal adverse effects related to study medications | Within 24 hours after delivery
  Occurrence of maternal side effects including diarrhea, shivering, headache, facial flushing, nausea, or vomiting following administration of study medications.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Albazee E, Alrashidi H, Laqwer R, Elmokid SR, Alghamdi WA, Almahmood H, AlGhareeb M, Alfertaj N, Alkandari DI, AlDabbous F, Alkanderi J, Al-Jundy H, Abu-Zaid A, Alomar O. Intravenous Carbetocin Versus Rectal Misoprostol for the Active Management of the Third Stage of Labor: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Cureus. 2022 Oct 12;14(10):e30229. doi: 10.7759/cureus.30229. eCollection 2022 Oct. PMID 36246091
- [Result] Delavallade M, Vaunois A, Cellier M, Boukerfa-Bennacer Y, Chauleur C, Raia-Barjat T. Carbetocin versus oxytocin for the prevention of postpartum haemorrhage during caesarean section in patients at high risk of bleeding. Eur J Obstet Gynecol Reprod Biol. 2024 Sep;300:206-210. doi: 10.1016/j.ejogrb.2024.07.015. Epub 2024 Jul 8. PMID 39029242
- [Result] Rath W. Prevention of postpartum haemorrhage with the oxytocin analogue carbetocin. Eur J Obstet Gynecol Reprod Biol. 2009 Nov;147(1):15-20. doi: 10.1016/j.ejogrb.2009.06.018. Epub 2009 Jul 17. PMID 19616358
- [Result] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571